CLINICAL TRIAL: NCT01871207
Title: Serum and Intraocular Levels of Erythropoietin and VEGF in Type 2 Diabetes Patients With Proliferative Retinopathy
Acronym: UVA-EVA
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Anna Cancarini, M.D., Università degli Studi di Brescia
Other Study IDs: UVA-EVA
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Diabetic Retinopathy
Keywords: Erythropoietin (EPO); Diabetes; Diabetic Retinopathy; Vascular Endothelial Growth Factor (VEGF); Erythropoiesis Stimulating Agents (ESA)
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic patients: Diabetic patients who underwent vitrectomy for Proliferative Diabetic Retinopathy
- Non-diabetic patients: Non-diabetic patients who underwent vitrectomy for macular hole or pucker

SUMMARY:
Some studies have recently shown that the concentration of erythropoietin in the vitreous humor of diabetic patients suffering from diabetic retinopathy is higher than non-diabetic patients. It was reported a higher concentration of erythropoietin in vitreous humor than blood, indicating a local production. In some cases it was also found a positive association between concentrations of Erythropoietin and Vascular Endothelial Growth Factor (VEGF). Both of these factors, erythropoietin and VEGF, show important angiogenic activity and may play a role in the development of diabetic retinopathy.

This study enrolled type 2 diabetic patients with PDR who had to undergo vitrectomy during the period May 2011-January 2012 at the Unit of Ophthalmology, A.O. Civil Hospital and University of Brescia. Inclusion criteria were the following: type 2 diabetes, age greater than 18 years, and PDR; exclusion criteria were: age less than 18 years, type 1 diabetes, initial DR, PDR patients not requiring surgery, previous vitrectomy in the eye under examination or other ophthalmic surgery or laser therapy within the previous 3 months.

Non-diabetic patients who underwent vitrectomy for macular hole or pucker represented the control group (CTRLs); their inclusion criteria were: age greater than 18 years and the presence of macular pucker or macular hole requiring vitrectomy. Exclusion criteria were: age less than 18 years, diagnosis of diabetes mellitus, and previous vitrectomy in the eye under examination or other ophthalmic surgery or laser therapy within the previous 3 months. All patients underwent a complete ophthalmologic examination (visual acuity, slit lamp, tonometry, fluorescein retinal angiography, and optical coherence tomography -OCT-). Informed consent was obtained from all patients after a detailed description of the aims and procedures of the study.

The following data were recorded for each patient:

1. Population: age (years), sex (M/F);
2. Clinical: diabetes (Absent or Type 2); time since initial diagnosis of diabetes (years); type of therapy for DM: diet, oral hypoglycaemic agents, mixed (oral agents and insulin, insulin); hypertension (defined as systolic blood pressure > 140 and diastolic blood pressure > 90 mmHg or on antihypertensive drugs); current (Yes/No) antihypertensive therapy; use of angiotensin II receptor blockers (ARB) or angiotensin converting enzyme inhibitors (ACE-i); presence of hypercholesterolaemia, comorbidities, therapy with statins (Yes/No), anticoagulants (Yes/No), antiplatelet therapy (Yes/No); other therapies performed, smoking (non-smoker, active smoker); complications of diabetes mellitus present at the time of evaluation (heart disease, nephropathy, neuropathy);
3. Ocular: eye (OD/OS); visual acuity; presence and grade of diabetic retinopathy; presence of emovitreo; presence of diabetic macular oedema; presence of cataract or lens implant; intervention with phacoemulsification during vitrectomy; presence of retinal diseases, or any other concomitant eye diseases; performance of previous retinal laser therapy, intravitreal injection of Avastin before the vitrectomy;
4. Biochemical: Haemoglobin (g/dL); glucose (mg/dL); glycated haemoglobin (%); platelets (N/mmc); creatinine (mg/dL); albuminuria (mg/day), creatinine clearance (mL/min), calculated by the Modification of Diet in Renal Disease (MDRD) formula; total cholesterol (mg/dL); HDL and LDL; triglycerides (mg/dL).

All patients underwent a 23- or 25-gauge pars plana vitrectomy. The primary outcome of the study was the measurement of EPO and VEGF concentrations in serum and vitreous and aqueous humor. Blood samples, taken before surgery, were centrifuged at 3000 rpm for 10 minutes to separate the serum fraction, which was stored at -80°C. Aqueous and vitreous humor were taken during the surgery and immediately frozen at -80°C. Both EPO and VEGF concentrations were measured in serum and vitreous humor; however, owing to the small amount of sample, only EPO concentrations were determined in aqueous humor. EPO was assayed by radioimmunoassay (Immulite EPO 200, Siemens), with the lowest detection limit of 1.0 mIU/mL. VEGF was assayed by ELISA (Human VEGF Immunoassay, R & D Systems Europe, Abingdon, UK) with a lower limit of detection of 10.0 pg/mL. VEGF concentrations below the lower limit of detection were set to 5 pg/mL to perform statistical analysis. VEGF values above 2000 pg/mL were set to 2500 pg/mL; statistical tests were also performed after deleting the data above 2000 pg/mL.

ELIGIBILITY:
CASE

Inclusion criteria:

* type 2 diabetes,
* age greater than 18 years, and
* PDR.

Exclusion criteria were:

* age less than 18 years,
* type 1 diabetes,
* initial DR,
* PDR patients not requiring surgery,
* previous vitrectomy in the eye under examination or other ophthalmic surgery or laser therapy within the previous 3 months.

CONTROL

Inclusion criteria:

* age greater than 18 years and the presence of macular pucker or macular hole requiring vitrectomy.

Exclusion criteria were:

* age less than 18 years,
* diagnosis of diabetes mellitus, and
* previous vitrectomy in the eye under examination or other ophthalmic surgery or laser therapy within the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case: type 2 diabetic patients with PDR who had to undergo vitrectomy during the period May 2011-January 2012 at the Unit of Ophthalmology, A.O. Civil Hospital and University of Brescia.
  Control: non-diabetic patients who underwent vitrectomy for macular hole or pucker.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Ocular concentration of Erythropoietin and VEGF. | eight months

CONTACTS AND LOCATIONS:
Locations (1):
- Spedali Civili di Brescia, Brescia, Brescia, Italy